CLINICAL TRIAL: NCT07146581
Title: Primary Care Screening and Intervention for Caregiving Assessment and Support for Patients With Dementia: Technology-Based Intervention Usability and Pilot Testing
Brief Title: Technology-Based Intervention Usability and Pilot Testing
Acronym: SIRENS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-05027492; R61AG079012 (NIH)
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Elder Abuse; Elder Neglect
Keywords: Older Adults; Technology
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: SIRENS Intervention (Experimental): The SIRENS intervention is a technology intervention designed specifically for caregivers of those with dementia, providing them with easy access to expert-reviewed information and helpful resources. The content includes take-home messages summarizing the main points discussed and a goal-setting feature that encourages the care givers to establish small, actionable goals.
  Interventions: Behavioral: SIRENS

INTERVENTIONS:
Behavioral: SIRENS — The SIRENS intervention is a technology intervention designed specifically for caregivers of those with dementia, providing them with easy access to expert-reviewed information and helpful resources. The content includes take-home messages summarizing the main points discussed and a goal-setting feature that encourages the care givers to establish small, actionable goals.

SUMMARY:
This research project has three main goals:

(1) To create a new screening tool that helps primary care doctors spot signs of neglect in older adults with dementia. (2) To design a support program that can be delivered both in person and through a mobile app on Android phones. (3) To run a clinical trial with three groups of participants to find out how effective the screening tool is on its own, and how effective it is when combined with the support program-compared to standard care.

This current phase of the project focuses on parts of goals 1 and 2, as described below.

DETAILED DESCRIPTION:
Elder abuse is common and has serious health consequences but is under-recognized and under-reported. Older adults with dementia are at much higher risk of mistreatment than other older adults, and the risk of mistreatment has been shown to be greater with increasing severity of dementia. This mistreatment is usually perpetrated by caregivers.

Screening for elder mistreatment and initiation of intervention in primary care clinics may be helpful, but few evidence-based tools or strategies exist. As few tools exist that may be effectively used in a busy clinical setting, evidence of the impact of screening and potential subsequent intervention on patient-important outcomes is lacking. Further, existing tools were developed for and studied in cognitively intact older adults and may not be appropriate for older adults with AD/ADRD.

In addition, elder mistreatment includes physical abuse, sexual abuse, verbal/emotional/psychological abuse, financial exploitation, and caregiver neglect. These different types of elder mistreatment represent very different phenomena, occur in various groups of older adults, and respond to very different intervention strategies. These discrepancies have made connecting positive identifications of mistreatment in the primary care setting to the next steps, including interventions, very challenging. Focusing on an intervention for caregiver neglect in older adults with dementia has the potential to address these challenges. Given that the severity of dementia represents a significant risk factor in the caregiving relationship, our goal is to provide support for dementia caregivers.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old or older
* Provides care for a patient at the Center on Aging who meets the following criteria:
* Patient is at least 65 years old
* Patient has diagnosed dementia
* Patient requires assistance with at least 1 ADL
* Self-identifies as primary informal caregiver for an older adult
* Provides at least 8 hours per week of direct care (may include logistics, oversight, observation, as well as hands-on care, but must include at least some in-person assistance)
* Can read and speak English at a 6th grade level or above
* Not blind or deaf
* No active plan to disengage from providing care to the older adult within the next year
* Ability to travel to the COA or CABR for study activities and/or attend study session(s) virtually through Zoom on their personal device

Exclusion Criteria:

* Non-fluent English speaker
* Hired caregiver
* Provides care for a patient in hospice care
* Too ill or weak to complete the interviews (per the interviewer)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-18 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived system feasibility, acceptability, and usability of the SIRENS intervention as measured by the Mean Difference in Score of the Program Evaluation Questionnaire. | 1 week post-intervention
  System feasibility, acceptability and usability will be assessed in the Program Evaluation Questionnaire. This is based on the Davis Perceived Usefulness, Perceived Ease of Use, and User Acceptance Scale. Response options range from 1= Strongly Disagree to 7= Strongly agree. Questions include those asking about the technology and components of the intervention. Total scores range from 23 to 161. Higher scores indicate greater user acceptance of the technology.
Perceived system feasibility, acceptability, and usability of the SIRENS intervention as measured by a qualitative interview assessment | 1-week post intervention
  System feasibility, acceptability and usability will be assessed in care partner participants using a semi-structured interview. Thematic analyses will be used to assess qualitative interviews.

SECONDARY OUTCOMES:
Mean difference in score of caregiver burden, as measured by the Zarit Caregiver Burden Assessment. | Baseline and 1 week post-intervention
  Caregiver burden will be assessed in care partner participants using the reliable and valid Zarit Caregiver Burden Assessment. Response options range from 0= Never to 4= Nearly always. Questions include those asking about relationship with the care recipient and stress. Overall scores range from 0 to 48, with higher scores indicating more caregiver burden.
Mean difference in score of caregiver quality of life, as measured by the Quality of Life Inventory | Baseline and 1 week post-intervention
  Caregiver quality of life will be assessed in care partner participants using the reliable and valid Quality of Life Inventory. Questions include those asking about importance (on a 3-point rating scale, higher value indicating more importance) and satisfaction (on a 6-point rating scale, higher value indicating more satisfaction) of life domains. Importance scores are multiplied by satisfaction scores for each domain, and then these scores are summed to determine the overall score. Overall scores range from -96 to 96, with higher scores indicating higher quality of life.
Mean difference in score of caregiver preparedness, as measured by the Caregiver Preparedness Scale | Baseline and 1 week post-intervention
  Caregiver preparedness will be assessed in care partner participants using the Preparedness Scale. Response options range from 0= Not at all prepared to 4= Very well prepared. Overall scores range from 0 to 24 with higher scores indicating more feelings of preparedness.
Mean difference in score of caregiving self-efficacy, as measured by the Caregiving Self-Efficacy Scale | Baseline and 1 week post-intervention
  Caregiving self-efficacy will be measured in care partner participants by a modified Caregiving Self-Efficacy Scale. Response options range from 0= Can not do at all to 100= Certainly can do. Overall scores range from 0 to 900 with higher scores indicating more confidence.
Mean difference in score of caregiver depression, as measured by the Center for Epidemiologic Studies Depression Scale | Baseline and 1 week post-intervention
  Caregiver depression will be assessed in care partner participants using the reliable and valid Center for Epidemiologic Studies Depression Scale. Response options range from 0= Rarely or none of the time to 3= Most or almost none of the time. Overall scores range from 0 to 60 with higher scores indicating greater depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Rosen, MD, Principal Investigator — Weill Cornell Medical College of Cornell University; Sara J Czaja, PhD, Principal Investigator — Weill Cornell Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan for resource sharing is based on the National Institutes of Health/National Institute on Aging (NIH/NIA) Data Sharing Policy. The investigators plan, consistent with the NIH goals of data sharing, is to promote use of the rich SIRENS database by the larger research community as this will further the impact of SIRENS and expand possibilities for collaboration. It will also allow other researchers to expedite the translation of the research findings into knowledge, products, and procedures. Further, the plan is devised to make the data as widely and freely available as possible while at the same time safeguarding the privacy of participants and protecting confidential and proprietary data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data from research projects will be made available no later than acceptance of publication of the main findings from the final data set. There is no end date to access the data from the research projects.
Access Criteria: The investigators agree to share the data with researchers working under an institution with Federal Wide Assurance who agree to a data sharing agreement that stipulates protection of participant privacy and data confidentiality, acknowledgement of SIRENS, that the data will be used for research purposes only, and that the data will not be transferred to other users. The computerized data will include raw data, derived variables, all necessary documentation as described in the National Archive of Computerized Data on Aging depositor agreement. All data will be de-identified. The investigators will follow the guides published by the US Department of Health and Human Services in this respect. Each data set will include data documentation to ensure that others can use the data set and to minimize confusion. Information about where and how to locate and access the data will be available in any publications and presentations authored by SIRENS investigators.